CLINICAL TRIAL: NCT07055282
Title: SGLT2i in Calcium Kidney Stones
Brief Title: SGLT2i in Kidney Stones
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0673; 1R01DK144310 (NIH)
Record Dates: First submitted 2025-06-24; First posted 2025-07-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones
Keywords: kidney stones; SGLT2i; empagliflozin; calcium kidney stones; kidney stone; calcium kidney stone
MeSH Terms: conditions — Kidney Calculi | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CaP (Calcium Phosphate) stone patients (Active Comparator): Defined as >50% calcium phosphate content on most recent stone analysis Age 18-70 years
  Interventions: Drug: Empagliflozin (Jardiance®)
- CaOx (Calcium Oxalate) stone patients (Active Comparator): Defined as >50% calcium oxalate content on most recent stone analysis Age 18-70 years
  Interventions: Drug: Empagliflozin (Jardiance®)

INTERVENTIONS:
Drug: Empagliflozin (Jardiance®) — Empagliflozin (Jardiance®), 10 mg tablet taken orally once daily for 4 weeks. Dispensed at baseline by the Investigational Drug Service. It will be administered at home by participants.

SUMMARY:
This study is looking at whether empagliflozin, a medication typically used for diabetes and heart conditions, may affect factors that contribute to kidney stone formation. The research focuses on people who have had calcium-based kidney stones, i.e. calcium oxalate or calcium phosphate stones.

Previous studies in those without kidney stones found that empagliflozin increased urinary citrate levels without raising urine pH. The investigators are testing whether similar effects occur in people with a history of kidney stones.

Participants will take empagliflozin daily for 4 weeks. The investigators will collect 24-hour urine samples before and after treatment to measure various factors that influence stone formation, including citrate levels, pH, and calculated stone formation risk. The investigators will enroll 32 participants: 16 with a history of calcium oxalate stones and 16 with calcium phosphate stones.

Results from this study may inform future larger clinical trials investigating empagliflozin as a kidney stone prevention strategy.

DETAILED DESCRIPTION:
This is a single-center, prospective pilot study designed to evaluate the effects of the sodium-glucose co-transporter 2 inhibitor (SGLT2i), empagliflozin, on urinary risk factors in individuals with recurrent idiopathic calcium phosphate (CaP) or calcium oxalate (CaOx) kidney stones. Although empagliflozin is FDA-approved for other indications, it is being used off-label in our study to explore its potential for kidney stone prevention. The investigators' goal is to assess changes in urinary parameters relevant to stone formation, including citrate excretion, pH, and other metabolic markers.

Eligible participants will be adults aged 18 to 70 years with a documented history of CaP or CaOx kidney stones. Participants will be asked to stop certain medications and supplements prior to and during the study period if deemed safe by their primary care provider or nephrologist.

Each participant will complete two in-person study visits at the University of Chicago Clinical Research Center (CRC), a special research clinic, over approximately 4 weeks. They will also collect two 24-hour urine samples-one before starting the study drug and one at the end of the study. In addition, participants will take empagliflozin 10 mg once daily during the 4-week period and complete a brief phone or video check-in around the 2-week mark.

Laboratory tests and physical measurements will be performed during each visit. All urine samples will be analyzed by a central clinical laboratory (Litholink), and select samples will be stored for future analysis. Participants will be compensated for completing the study.

This pilot study is not intended to support a new drug indication or FDA labeling change. The findings will inform the design of a larger, hypothesis-driven study on the use of SGLT2 inhibitors in kidney stone prevention.

ELIGIBILITY:
Inclusion Criteria:

Calcium phosphate (CaP) stone participants:

* Age 18-70
* History of at least one calcium phosphate (hydroxyapatite) stone

  * Defined as at least 50% of stone material on most recent stone analysis

Calcium oxalate (CaOx) stone participants:

* Age 18-70
* History of at least one calcium oxalate stone

  * Defined as at least 50% of stone material on most recent stone analysis.

Other inclusion criteria considerations: The investigators will study balanced numbers of male and females. Prior studies did not have balanced representation of male and female sexes. In prior studies, less than 40% were female, or sex data is not presented. Study of both male and female sex is crucial with kidney stones and therapies that affect citrate and pH because there are well established epidemiologic differences in stone type and physiologic differences in acid-base handling by sex. Epidemiologically, younger women are more likely to have CaP stones, and this is likely because they have higher urine pH.

Exclusion Criteria:

* History of primarily brushite, uric acid, cysteine, or struvite stones
* History of severe acid-base abnormality, very low (less than 100mg/day) or very high (greater than 1500mg/day) urine citrate
* Participants who cannot stop diuretic medication or alkali supplementation for the course of the study period
* Use of drugs that can directly affect proximal tubule function (e.g., topiramate)
* Diagnosis of complete distal renal tubular acidosis
* Diagnosis of chronic kidney disease (eGFR <60 mL/min/1.73m²)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in calcium phosphate | 4 weeks
  Calcium phosphate supersaturation will be measured or calculated at baseline and study completion. The investigators will calculate change in calcium phosphate supersaturation for all participants and within each group.
Change in urine citrate | 4 weeks
  Urine citrate will be measured or calculated at baseline and study completion. The investigators will calculate change in urine citrate for all participants and within each group.
Change in pH | 4 weeks
  pH will be measured or calculated at baseline and study completion. The investigators will calculate change in pH for all participants and within each group.
Calcium oxalate supersaturation | 4 weeks
  Calcium oxalate supersaturation will be measured or calculated at baseline and study completion. The investigators will calculate change in calcium oxalate supersaturation for all participants and within each group.

SECONDARY OUTCOMES:
Change in 24-hour urine citrate excretion (mg/day) from baseline to 4 weeks | 4 weeks
  24-hour urine citrate excretion will be measured at baseline and study completion. The change from baseline to 4 weeks will be calculated for each participant and compared between CaP and CaOx stone groups.
Change in urine pH from baseline to 4 weeks | 4 weeks
  Urine pH will be measured at baseline and study completion. The change from baseline to 4 weeks will be calculated for each participant and compared between groups.
Change in calcium phosphate supersaturation from baseline to 4 weeks | 4 weeks
  Calcium phosphate supersaturation will be calculated using EQUIL2 at baseline and 4 weeks. The change will be calculated for each participant and compared between groups.
Change in calcium oxalate supersaturation from baseline to 4 weeks | 4 weeks
  Calcium oxalate supersaturation will be calculated using EQUIL2 at baseline and 4 weeks. The change will be calculated for each participant and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States